CLINICAL TRIAL: NCT02152943
Title: Combination Treatment With Everolimus, Letrozole and Trastuzumab in Hormone Receptor and HER2/Neu-Positive Patients With Advanced Metastatic Breast Cancer and Other Solid Tumors: Evaluating Synergy and Overcoming Resistance
Brief Title: Everolimus, Letrozole and Trastuzumab in HR- and HER2/Neu-positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0119; NCI-2014-01615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0119 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Advanced Malignant Solid Neoplasm; Estrogen Receptor Positive; HER2/Neu Positive; Postmenopausal; Premenopausal; Progesterone Receptor Positive; Recurrent Breast Carcinoma; Refractory Breast Carcinoma; Refractory Hormone Receptor Positive Breast Carcinoma; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Letrozole; Trastuzumab; PF-05280014; Ogivri; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (everolimus, letrozole, trastuzumab) (Experimental): Patients receive everolimus PO QD and letrozole PO QD. Patients also receive trastuzumab IV over 30-90 minutes once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Biological: Trastuzumab

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab-dkst

SUMMARY:
This phase I trial studies the side effects and best dose of everolimus and trastuzumab when given together with letrozole in treating patients with hormone receptor-positive and human epidermal growth factor (EGF) receptor 2 (HER2)-positive breast cancer or other solid tumors that have spread to other places in the body. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by blocking the use of estrogen by tumor cells. Immunotherapy with monoclonal antibodies, such as trastuzumab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving everolimus, letrozole, and trastuzumab together may be a better treatment for breast cancer and other solid tumors than everolimus alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine reasonable dose of drugs in treatment combination, including maximum tolerated dose (MTD) and toxicity profiles, via a brief initial "run-in"/dose escalation.

II. Evaluate response, in patients with tumors that demonstrate hormone receptor (HR)-positivity (> 1% on immunohistochemistry [IHC]) and human EGF receptor 2 (HER)-positivity (IHC 3 and/or IHC 2/3 and fluorescence in situ hybridization [FISH] amplification).

SECONDARY OBJECTIVES:

I. Correlate activity of combination with genomic and proteomic signatures. II. Evaluate 2 expanded cohorts of patients to include: 1) HR- and HER2-positive breast cancer (n=12) and 2) other HR- and HER2-positive tumors that have demonstrated activity in the dose escalation portion of the study (n=12).

OUTLINE: This is a dose-escalation study of everolimus and trastuzumab.

Patients receive everolimus orally (PO) once daily (QD) and letrozole PO QD. Patients also receive trastuzumab intravenously (IV) over 30-90 minutes once every 3 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to any screening procedures
* Performance status =< 1
* Absolute neutrophil count (ANC) >= 1 x 10^9/L
* Platelets >= 75 x 10^9/L
* Hemoglobin (Hb) > 8 g/dL
* Total serum bilirubin =< 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN in patients with liver metastases)
* International normalized ratio (INR) =< 2
* Serum creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL or =< 7.75 mmol/L and fasting triglycerides =< 2.5 x ULN; Note: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Histologically confirmed advanced solid tumors with HR-positivity defined as > 1% on immunohistochemistry (estrogen receptor-positive with or without positivity for the progesterone receptor) and HER2/neu positivity (3+ on IHC and/or 2+ on IHC and FISH amplified, or by v-erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 [ERBB2] mutation on next generation sequencing)
* Must have measurable or evaluable disease
* At least 4 weeks since the last dose of chemotherapy, immunotherapy, surgery, or radiation therapy (exception: patients may have received palliative low dose radiation therapy one week before treatment provided it is not given to the only targeted lesions); at least 6 weeks for therapy which is known to have delayed toxicity (nitrosoureas, mitomycin-C, and liposomal doxorubicin); at least 4 weeks (or 5 half-lives, whichever is shorter) since treatment with biologic/targeted therapies; at least 2 weeks since last hormonal therapy
* Female patients must either be: post-menopausal women as defined by a) age >= 60 years of age; b) prior bilateral oophorectomy; c) age < 60 with at least 12 months of spontaneous amenorrhea or post-menopausal range follicle stimulating hormone (FSH) and estradiol levels or premenopausal women receiving a gonadotropin-releasing hormone agonist
* Patient may have had any number of prior chemotherapy regimens in the adjuvant/neoadjuvant and/or metastatic setting (including none)
* Patient may have had any number of prior treatments with anti-HER2 strategies in the adjuvant/neoadjuvant and/or metastatic setting (including none)
* Patient may have had any number of prior hormonal therapies in the adjuvant/neoadjuvant and/or metastatic setting (including none)
* Breast cancer patients in the expansion cohort must be hormone sensitive or have refractory disease

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by glycated hemoglobin (HbA1c) > 8% despite adequate therapy; patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Patients who have any severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction 6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Symptomatic congestive heart failure of New York Heart Association class III or IV
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA])
  * Known severely impaired lung function (spirometry and diffusion capacity of the lungs for carbon monoxide [DLCO] 50% or less of normal and oxygen [O2] saturation 88% or less at rest on room air)
  * Active, bleeding diathesis
* Chronic treatment with corticosteroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed
* Known history of human immunodeficiency virus (HIV) seropositivity
* Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study; patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, bacillus Calmette-Guérin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Patients who have a history of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for >= 3 years
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after; highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository
  * Total abstinence or
  * Male/female sterilization
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* History of allergic reactions or hypersensitivity to compounds similar to trastuzumab and/or letrozole
* Left ventricular ejection fraction (LVEF) < 50%
* Patients with corrected QT (QTc) interval > 0.47 seconds
* Prior exposure to more than 360 mg/m^2 doxorubicin, more than 120 mg/m^2 mitoxantrone, or more than 90 mg/m^2 idarubicin, or elevated baseline cardiac troponin I
* Drugs with potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and inducers should be avoided during the course of treatment
* Patients with active central nervous system (CNS) metastasis and/or carcinomatous meningitis; however, patients with CNS metastasis (except leptomeningeal disease) who have completed a therapy and are clinically stable for 3 weeks as defined as: (1) no evidence of new or enlarging CNS metastasis and (2) off steroids and/or anticonvulsants may be eligible
* Patient is known to be hepatitis B or hepatitis C-positive (these tests are not required)
* Patients with current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and/or recommended phase II dose | 21 days
  Defined as the highest dose at which no more than 1 of 6 patients has had dose-limiting toxicity.
Clinical benefit rate | Up to 4 years
  Defined as the percentage of patients with stable disease >= 6 months/partial response/complete response. The point estimate and the 90% exact confidence interval for the clinical benefit rate will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Ballhausen A, Wheler JJ, Karp DD, Piha-Paul SA, Fu S, Pant S, Tsimberidou AM, Hong DS, Subbiah V, Holley VR, Huang HJ, Brewster AM, Koenig KB, Ibrahim NK, Meric-Bernstam F, Janku F. Phase I Study of Everolimus, Letrozole, and Trastuzumab in Patients with Hormone Receptor-positive Metastatic Breast Cancer or Other Solid Tumors. Clin Cancer Res. 2021 Mar 1;27(5):1247-1255. doi: 10.1158/1078-0432.CCR-20-2878. Epub 2020 Oct 28. PMID 33115815
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org